CLINICAL TRIAL: NCT03432442
Title: Pharmacokinetics and Pharmacodynamics of Ivermectin in Pediatric Dengue Patients
Acronym: PKIDEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIR17003
Record Dates: First submitted 2017-12-21; First posted 2018-02-14 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Dengue Hemorrhagic Fever
MeSH Terms: conditions — Severe Dengue | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (6 dengue patients) (Experimental): Volunteers weighed > 30 kg receiving 400 µg of ivermectin per 1 kg of body weight
  Interventions: Drug: Ivermectin
- Group 2 (6 dengue patients) (Experimental): Volunteers weighed 15 to 30 kg receiving 400 µg of ivermectin per 1 kg of body weight
  Interventions: Drug: Ivermectin
- Group 3 (6 dengue patients) (Experimental): Volunteers weighed > 30 kg receiving 600 µg of ivermectin per 1 kg of body weight
  Interventions: Drug: Ivermectin
- Group 4 (6 dengue patients) (Experimental): Volunteers weighed 15 to 30 kg receiving 600 µg of ivermectin per 1 kg of body weight
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Ivermectin once every 24 hours for three administrations

SUMMARY:
Design and Outcomes This research study is designed as open-label, sequential dose-escalating clinical trial. There will be two phases of enrollment.

In the first phase, pediatric dengue patients with body weight greater than 30 kg will be recruited. The first six volunteers will be administered with 400 μg/kg every 24 hours for a total of three times. The last six volunteers will be administered with 600 μg/kg every 24 hours for a total of three times.

In the second phase, pediatric dengue patients with body weight between 15 to 30 kg will be recruited. Similar to the first phase, the first six and the last six volunteers will be administered with 400 μg/kg and 600 μg/kg every 24 hours for a total of three times, respectively.

A total of 24 volunteers will be recruited from Faculty of Medicine Siriraj hospitals

DETAILED DESCRIPTION:
The research team has planned to conduct three interim analyses for safety and one final report. The interim analyses will be conducted as follows:

1. First interim analysis: After the completion of the last volunteer of the group with body weight >30 kg receiving ivermectin 400 μg/kg every 24 hours for a total of three times (i.e. the sixth volunteer).
2. Second interim analysis: After the completion of the last volunteer of the group with body weight >30 kg receiving ivermectin 600 μg/kg every 24 hours for a total of three times (i.e. the twelfth volunteer).
3. Third interim analysis: After the completion of the last volunteer of the group with body weight 15 to 30 kg receiving ivermectin 400 μg/kg every 24 hours for a total of three times (i.e. the twelfth volunteer).

The results of each interim analyses will be submitted to DSMB to determine whether the study is safe to be conducted in the next group of volunteers. Additionally, the results of interim analyses and the safety assessments from DSMB will be submitted to all ECs

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 1-15 years 0 day
2. Weight is equal or greater than 15 kg
3. History or presence of acute fever within the last 72 hours diagnosed as acute dengue virus infection
4. Patients who are expected to be able to start the study drug within 72 hours of fever
5. Written informed consent to enroll in the study is obtained from parents or legal representatives and/or patients.
6. The test for dengue nonstructural protein 1 is positive, or PCR screening for viral genome is positive
7. Female patients with history of menarche need to have a negative result for urine pregnancy test, except during a menstrual period.

Exclusion Criteria:

1. Has significant underlying disease(s) that can affect the study outcome or the study participation may be harmful to patients with those underlying diseases including but not limited to:

   * Kidney disease
   * Thalassemia
   * congenital heart disease
   * epilepsy
   * cerebral palsy Other underlying diseases may result in exclusion depending on the judgement of investigator.
2. Having developed or showed the following laboratory values, warning signs or signs of severe dengue including:

   * AST and/or ALT levels > 500 IU/L
   * Platelets count < 50,000 cells/mm3
   * Abdominal pain or tenderness
   * Persistent vomiting
   * Clinical fluid accumulation such as pleural effusion, ascites
   * Mucosal bleeding
   * Lethargy/restlessness
   * Liver enlargement >2 cm
   * Increase in Hct concurrent with rapid decrease in platelet count
   * Severe plasma leakage such as dengue shock syndrome, fluid accumulation with respiratory distress
   * Severe bleeding as evaluated by clinician
   * Severe organ involvement including but not limited to acute liver failure, altered level of consciousness (e.g. encephalopathy, encephalitis), seizure or other CNS unusual manifestation, acute renal failure, cardiomyopathy and other unusual manifestation
3. History of ivermectin allergy or receiving medications that increase gamma-aminobutyric acid (GABA) potentiating activity such as barbiturates, benzodiazepines, sodium oxybate, valproic acid, or receiving medications that prevent p-glycoprotein transport system such as amiodarone, carvedilol, clarithromycin, cyclosporine, erythromycin, itraconazole, ketoconazole, quinidine, ritonavir, tamoxifen, verapamil, amprenavir, clotrimazole, phenothiazines, rifampin, St. John's Wort etc.
4. Currently receiving immunosuppressive agents such as steroid (except topical steroid), chemotherapeutic agents or have discontinued these medications for less than a month
5. Having a history of receiving ivermectin within one month
6. Inability to ingest medications in a form of tablets as informed by patients and their parents or legal representatives

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ivermectin in pediatric dengue patients | 7 days
  Blood samples will be collected, and ivermectin plasma concentrations will be measured with High Performance Liquid Chromatography-Tandem Mass Spectrometry (HPLC-MS/MS).

SECONDARY OUTCOMES:
Pharmacodynamic effects of ivermectin on viral load in plasma of pediatric dengue patients | 7 days
  Blood samples will be collected, and viral load in plasma will be measured with quantitative RT-PCR.
Pharmacodynamic effects of ivermectin on NS1 antigen in plasma of pediatric dengue patients | 7 days
  Blood samples will be collected, and NS1 antigen in plasma will be measured with NS1-ELISA assay.
Viremia clearance | 7 days
  Time between the first drug administration and the point of specimen collection at which viral load becomes undetectable
NS1 antigenemia clearance | 7 days
  Time between the first drug administration and the point of specimen collection at which NS1 antigen becomes undetectable
Occurrences of adverse events | 7 days
  The number of volunteers with any adverse events by the total number of volunteers in the treatment group
Occurrences of abnormal laboratory result | 7 days
  The number of volunteers with any change of laboratory results from normal at baseline to abnormal during the study by the total number of volunteers in the treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Panisadee Avirutnan, Assoc. Prof., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Tropical Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided